CLINICAL TRIAL: NCT03668431
Title: A Phase 2 Study of Dabrafenib and Trametinib in Combination With PDR001 in Patients With BRAFV600E Metastatic Colorectal Cancer
Brief Title: Dabrafenib + Trametinib + PDR001 In Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Novartis (Industry); Stand Up To Cancer (Other)
Responsible Party: Principal Investigator, Ryan B Corcoran, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-144
Record Dates: First submitted 2018-09-11; First posted 2018-09-12 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — dabrafenib; trametinib; spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PDR001, Dabrafenib, Trametinib (Experimental): Patients who fulfill eligibility criteria will be entered into the trial to receive PDR001, Dabrafenib, Trametinib. Treatment will be administered on an outpatient basis.
  After the screening procedures confirm participation in the research study:
  * Dabrafenib will be taken twice a day for 28 consecutive days
  * Trametinib will be taken once a day for 28 consecutive days
  * PDR001 will be administered IV every 28 days.
  Interventions: Drug: Dabrafenib; Drug: Trametinib; Drug: PDR001

INTERVENTIONS:
Drug: Dabrafenib — Dabrafenib will be taken twice a day for 28 consecutive days
  .
  Other Names: Tafinlar®
Drug: Trametinib — Trametinib will be taken once a day for 28 consecutive days
  Other Names: Mekinist®
Drug: PDR001 — PDR001 will be administered IV every 28 days

SUMMARY:
This research study is studying a combination of drugs as a possible treatment for metastatic colorectal cancer characterized by BRAF V600E mutation.

The names of the study drugs involved in this study are:

* Dabrafenib
* Trametinib
* PDR001

DETAILED DESCRIPTION:
* This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug combination to learn whether the drug combination works in treating a specific disease. "Investigational" means that the drug combination is being studied.

  * The FDA (the U.S. Food and Drug Administration) has not approved PDR001 as a treatment for any disease.
  * The FDA has not approved dabrafenib and trametinib for your specific disease but it has been approved for other uses, whether alone as single agents, or given together as in this study.
* This research study is studying a combination of drugs as a possible treatment for metastatic colorectal cancer characterized by BRAF V600E mutation.

  * All humans have a gene called BRAF which is responsible for sending signals to proteins called B-Raf inside of cells that help them grow. In some metastatic colorectal patients, this gene mutates and causes cancer cells to grow in uncontrolled ways.

    --- Dabrafenib is a drug that is thought to inhibit the mutant BRAF activity, which may serve to slow or stop cell growth of metastatic colon cancer.
  * Mitogen-activated protein kinase (MAPK) is a pathway that helps to activate the BRAF mutated genes. The MAPK pathway is commonly found to be overactivated in BRAF mutated tumor cells. MEK (which refers to MAPK/ERK Kinase) enzymes are essential to the activity of the MAPK pathway.

    * Trametinib inhibits the MEK enzymes in order to shut down the MAPK pathway, thus blocking the pathway that helps the cancer cells grow uncontrollably.
    * PDR001 is a drug which binds to PD1 on immune cells and is believed to block binding of PD-L1 and PD-L2. PD-L1/PDL1 and PD-L2/PDL2 are often used by cancer cells and to escape the power of the body's immune system so that they cannot be fought. By blocking that binding of the molecules, the body's immune system may reach and fight the cancer cells. Researchers are hoping that administration of all three of these drugs may help anti-cancer activities work together to slow or stop the cancer growth and may help your own immune system damage or destroy the existing cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed metastatic colorectal cancer and a documented BRAF V600E mutation by a CLIA-certified laboratory test and must be wild-type for KRAS and NRAS.
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm with conventional techniques or as ≥10 mm with spiral CT scan, MRI, or calipers by clinical exam. See Section 11 for the evaluation of measurable disease.
* Patients may have received prior chemotherapy, prior anti-EGFR therapy, prior BRAF or MEK inhibitor, or prior immunotherapy (e.g. anti-PD1/PD-L1). Patients will also be allowed without prior treatments. If patient has been treated in the past, they must be at least 4 weeks since prior chemotherapy or radiation therapy.
* Age ≥ 18 years
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A)
* Life expectancy of greater than 3 months
* Participants must have normal organ and marrow function as defined below:

  * leukocytes ≥3,000/mcL
  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
  * creatinine within normal institutional limits --- OR
* creatinine clearance ≥ 60 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.

  * PT/INR <1.5 x ULN and PTT <1.5 ULN
  * Albumin > 2.5 g/dl
  * Patients must meet eligibility criteria on C1D1.
* LVEF > LLN by ECHO or MUGA
* The effects of trametinib, dabrafenib and PDR001 on the developing human fetus are unknown. For this reason and because these agents may be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of treatment.
* Ability to understand and the willingness to sign a written informed consent document.
* Subjects must avoid consumption of grapefruit, Seville oranges or products containing the juice of each during the entire study and preferably 7 days before the first dose of study medications, due to potential CYP3A4 interaction with the study medications. Orange juice is allowed.
* Exclusion Criteria
* Participants who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Participants who are receiving any other investigational agents.
* Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to of trametinib, dabrafenib or PDR001.
* Participants receiving any medications or substances that are strong inhibitors or inducers of CYP3A4 are ineligible but once on treatment must be used with caution. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list such as http://medicine.iupui.edu/clinpharm/ddis/table.aspx; medical reference texts such as the Physicians' Desk Reference may also provide this information. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because trametinib, dabrafenib or PDR001 have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with trametinib, dabrafenib or PDR001 breastfeeding should be discontinued if the mother is treated with trametinib, dabrafenib or PDR001.
* HIV-positive participants on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with trametinib, dabrafenib or PDR001. In addition, these participants are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.
* Active known or suspected autoimmune disease or a documented history of autoimmune disease, including ulcerative colitis and Crohn's disease (Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll).
* Systemic chronic steroid therapy (≥ 10mg/day prednisone or equivalent) or any immunosuppressive therapy 7 days prior to planned date for first dose of study treatment. Topical, inhaled, nasal and ophthalmic steroids are allowed.
* Current pneumonitis or interstitial lung disease.
* History of organ transplant requiring use of immunosuppressive medication.
* Taken an investigational drug ≤ 28 days or ≤ 5 half-lives (minimum 14 days) prior to start of study treatment, whichever is shorter.
* Current use of a prohibited medication.
* Malignant disease, other than that being treated in this study. Exceptions to this exclusion include the following: malignancies that were treated curatively and have not recurred within 2 years prior to study treatment; completely resected basal cell and squamous cell skin cancers and any completely resected carcinoma in situ.
* Active infection requiring systemic antibiotic therapy within 2 weeks prior to start of study treatment.
* Subjects with active Hepatitis B infection (HbsAg positive) will be excluded. Note: Subjects with antecedent of Hepatitis B (anti-HBc positive, HbsAg and HBV-DNA negative) are eligible.
* Subjects with positive test for hepatitis C ribonucleic acid (HCV RNA) Note: Subjects in whom HCV infection resolved spontaneously (positive HCV antibodies without detectable HCV-RNA) or those that achieved a sustained virological response after antiviral treatment and show absence of detectable HCV RNA ≥ 6 months (with the use of IFN-free regimes) or ≥ 12 months (with the use of IFN-based regimes) after cessation of antiviral treatment are eligible.
* Any medical condition that would, in the investigator's judgment, prevent the subject's participation in the clinical study due to safety concerns, compliance with clinical study procedures or interpretation of study results.
* Use of any live vaccines against infectious diseases within 4 weeks of initiation of study treatment
* Uncorrectable electrolyte abnormalities (e.g., hypokalemia, hypomagnesemia, hypocalcemia), long QT syndrome or taking medicinal products known to prolong the QT interval
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study treatments, their excipients, and/or dimethyl sulfoxide (DMSO).
* A history or current evidence/risk of retinal vein occlusion (RVO) or central serous retinopathy including:

  * Presence of predisposing factors to RVO or central serous retinopathy (e.g., uncontrolled glaucoma or ocular hypertension, uncontrolled hypertension, uncontrolled diabetes mellitus, or a history of hyperviscosity or hypercoagulability syndromes); or
  * Visible retinal pathology as assessed by ophthalmic examination that is considered a risk factor for RVO or central serous retinopathy such as:
  * Evidence of new optic disc cupping;
  * Evidence of new visual field defects on automated perimetry;
  * Intraocular pressure >21 mmHg as measured by tonometry.
* Cardiac or cardiac repolarization abnormality, including any of the following:

  * History or current diagnosis of cardiac disease indicating significant risk of safety for subjects participating in the study such as uncontrolled or significant cardiac disease, including any of the following:

    * Recent (within last 6 months) myocardial infarction (MI)
    * Unstable angina (within last 6 months),
    * Uncontrolled congestive heart failure (CHF)
    * Clinically significant (symptomatic) cardiac arrhythmias (e.g., sustained ventricular tachycardia, and clinically significant second or third degree atrioventricular [AV] block without a pacemaker).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-10-15 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | From the start of the treatment until disease progression/recurrence, up to approximately 5 years
  The participants best overall response will be assessed using RECIST 1.1 criteria
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  * Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
  * Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Number of participants with grade 3, 4 and 5 adverse events | From the start of treatment until 30 days after the last dose of a study drug, up to approximately 5 years
  Adverse Events will be assessed using Common Terminology Criteria for Adverse Events (CTCAE 4)

SECONDARY OUTCOMES:
Progression Free Survival | From the date of randomization until disease progression or death due to any cause, up to approximately 5 years
  Progression free survival is measured from the date of randomization/start of treatment to the date of event defined as the first documented progression or death due to any cause. Progression will be assessed using RECIST 1.1 Criteria.
  Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
Disease Control Rate | From the start of the treatment until disease progression/recurrence, up to approximately 5 years
  The number of participants that achieve either a Complete Response (CR), Partial Response (PR), or Stable Disease (SD) per RECIST 1.1 Criteria.
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  * Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Duration of Response | From the first documented response until the time of disease progression, up to approximately 5 years
  The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started, or death due to any cause. Participants without events reported are censored at the last disease evaluation). Response is assessed using RECIST 1.1 Criteria.
Overall Survival | From the date of randomization until the time of death, up to approximately 10 years
  Overall Survival (OS) is defined as the time from randomization (or registration) to death due to any cause, or censored at date last known alive.
Mechanisms of response and resistance to dabrafenib, trametinib, and PDR001 | Pre treatment and day 15
  Using multiplexed immune IF and RNAseq, assess the change in immune microenvironment between pre-treatment and day 15 on-treatment biopsies Using serial cfDNA analyses, monitor response and define mechanisms of resistance to this therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Corcoran, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hosital Cancer Center, Boston, Massachusetts
  - Dana Farber Cancer Institite, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tian J, Chen JH, Chao SX, Pelka K, Giannakis M, Hess J, Burke K, Jorgji V, Sindurakar P, Braverman J, Mehta A, Oka T, Huang M, Lieb D, Spurrell M, Allen JN, Abrams TA, Clark JW, Enzinger AC, Enzinger PC, Klempner SJ, McCleary NJ, Meyerhardt JA, Ryan DP, Yurgelun MB, Kanter K, Van Seventer EE, Baiev I, Chi G, Jarnagin J, Bradford WB, Wong E, Michel AG, Fetter IJ, Siravegna G, Gemma AJ, Sharpe A, Demehri S, Leary R, Campbell CD, Yilmaz O, Getz GA, Parikh AR, Hacohen N, Corcoran RB. Combined PD-1, BRAF and MEK inhibition in BRAFV600E colorectal cancer: a phase 2 trial. Nat Med. 2023 Feb;29(2):458-466. doi: 10.1038/s41591-022-02181-8. Epub 2023 Jan 26. PMID 36702949